CLINICAL TRIAL: NCT05903417
Title: A Randomised Open-Label Controlled Trial of Pleural Irrigation With Normal Saline Versus Intrapleural Tissue Plasminogen Activator and DNase (Fibrinolytic Therapy) in Pleural Infection.
Brief Title: Pleural Irrigation With Normal Saline Versus Intrapleural Fibrinolytic
Acronym: PENTAD-FT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2023-163
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Pleural Infection
MeSH Terms: interventions — Tissue Plasminogen Activator; dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleural Irrigation Arm (Active Comparator): subjects were administered 250 ml of 0.9% sodium chloride via chest tube a three way tap from a drip stand which were allowed drainage freely over 1 hour. Pleural irrigation will be performed minimum of 3 installations and maximum of 9 installation (3 times per day).
  Interventions: Other: Saline irrigation with 250 mls normal saline (over 1 hour)
- Intrapleural fibrinolytic arm (Active Comparator): t-PA (Alteplase) 5mg and DNase (Pulmozyme)5mg t-PA (Alteplase) that is available in our pharmacy is 50mg ampoule and DNase (Pulmozyme) is 2.5mg per ampoule The number of installation of intrapleural t-PA/DNase depends on the discretion of the treating physician (at least 6 hours apart between each dose). 5mg of Alteplase (t-PA) and 5mg DNase are diluted in each 50ml of 0.9% sodium.
  Both medication are administered sequentially which t-PA is first instilled intrapleurally and the chest tube is then clamped for 45 minutes, then unclamped to allow free drainage for 45 minutes. The same procedure is then repeated for DNase. Selection of the timing of treatment and removal of chest tube are depending on the chest physician's judgement.
  Interventions: Drug: Intrapleural fibrinolytic with alteplase 5mg and pulmozyme 5 mg

INTERVENTIONS:
Drug: Intrapleural fibrinolytic with alteplase 5mg and pulmozyme 5 mg — The number of installation of intrapleural t-PA/DNase depends on the discretion of the treating physician (at least 6 hours apart between each dose). 5mg of Alteplase (t-PA) and 5mg DNase are diluted in each 50ml of 0.9% sodium chloride solution. t-PA and DNase are not mixed together in one syringe. In brief , both medication are administered sequentially which t-PA is first instilled intrapleurally and the chest tube is then clamped for 45 minutes, then unclamped to allow free drainage for 45 minutes. The same procedure is then repeated for DNase. Selection of the timing of treatment and removal of chest tube are depending on the chest physician's judgement.
  Arms: Intrapleural fibrinolytic arm
Other: Saline irrigation with 250 mls normal saline (over 1 hour) — subjects were administered 250 ml of 0.9% sodium chloride via chest tube a three way tap from a drip stand which were allowed drainage freely over 1 hour. Pleural irrigation will be performed minimum of 3 installations and maximum of 9 installation (3 times per day).
  Arms: Pleural Irrigation Arm

SUMMARY:
Parapneumonic effusions caused by an infection of the pleural membranes occur in 40-57% of cases of pneumonia. A variable percentage (10-20%) of parapneumonic effusions progresses to empyema (pus) and/or abscess formation (encapsulation). Pleural infection is associated with significant morbidity and mortality which may be as high as 20-35% in immunocompromised patients Standard treatment of these collections in adults involves antibiotic therapy, effective drainage of infected fluid and surgical intervention if conservative management fails. For parapneumonic effusions which require clearance, appropriate therapy is effective drainage via an intercostal catheter (ICC) with antibiotic therapy. The presence of fibrinous septae in the pleural space, known as loculations, may result in inadequate drainage of effusions and therefore non-resolution of infection and systemic sepsis. Without effective intercostal catheter drainage, surgical intervention (VATS or open) has usually been required to clear loculations for resolution of infection.

Non-surgical treatment options to reduce the impact of adhesions and locule include (in addition to appropriate antibiotic therapy) single and multiple thoracocentesis, or single and multiple intercostal tube thoracostomies, with or without intrapleural fibrinolytic agents.

Fibrinolytic agents including streptokinase, urokinase, alteplase and recombinant tissue plasminogen activator (rTPA) have been used safely and effectively intrapleurally for complicated pleural effusion and empyema.

MIST 2 trial has established intrapleural therapy as the mainstay of CPEE treatment hence avoiding surgery and decreasing the length of hospitalization; however, little is known about the correct dosage needed for tPA and DNase. Dose and duration of intrapleural therapy based on MIST 2 involve multiple dosing and can be time-consuming for health care providers . Previous studies showed that complexity of treatment is a factor associated with poor adherence to a regimen. For this reason, trying to find the minimum effective dose and simplifying the regimen is essential for minimizing side effects and maximizing adherence. The review of currently available literature shows concurrent administration of tPA and DNase to be safe and effective even at lower cumulative dose Other study was carried out in May 2022 in which Modified regimen intrapleural alteplase 16 mg t-PA with 5 mg DNase for total 3 doses that administered sequentially within 24 h had been used. In this study, modified regimen of t-PA and DNase offer an alternative therapeutic option for patients that are unfit or refuse surgical intervention but persistent pleural infection. They have demonstrated similar treatment success comparable to other studies, as evidenced by improvement on pleural fluid drainage and reduction in pleural opacity on day 7 chest x-ray was approximately 50% from the baseline using intrapleural 16 mg t-PA with 5 mg DNase. The mechanism of action of t-PA and DNase in pleural cavity remain unclear. Studies suggested that IPFT may trigger the monocyte chemoattractant protein 1 (MCP-1) pathway which promote pleural fluid formation and subsequently causes a therapeutic lavage effect that increases pleural fluid drainage.

Another option for intrapleural therapy may be pleural irrigation with normal saline. The idea behind is to dilute and remove bacteria, cytokines, inflammatory cells, and pro-fibrinogenic coagulation factors, which induce pleural fluid organization. Also, the mechanical process of irrigation increases pleural fluid drainage by reducing stasis and organization of the intrapleural contents .

A randomised controlled pilot study in which saline pleural irrigation (three times per day for 3 days) plus best-practice management was compared with best-practice management alone was performed in patients with pleural infection requiring chest-tube drainage. The primary outcome was percentage change in computed tomography pleural fluid volume from day 0 to day 3. Patients receiving saline irrigation had a significantly greater reduction in pleural collection volume on computed tomography compared to those receiving standard care. Significantly fewer patients in the irrigation group were referred for surgery (30).

However, till date there is no study done on head to head comparison between intrapleural fibrinolytic with alteplase and DNAse Versus Pleural irrigationwith normal saline.

DETAILED DESCRIPTION:
Problem Statement

Retained complicated pleural effusion is associated with a risk of empyema and sepsis.IPFT is commonly used as the bridging therapy to surgery. The efficacy of saline irrigation is not known. However, the probable problem in this study is when failed saline irrigation, the patient will be given IPFT as part of the intention to treat.

Research Questions:

• Is the combination of intrapleural Alteplase (t-PA) 5mg and DNase (Pulmozyme) 5mg superior than pleural pleural irrigation in the management of pleural infection?

Primary Objective:

• To measure the volume of pleural effusion drainage (in mls) 48 hours following randomization

Secondary Objectives:

* To determine the reduction of pleural opacity (in percentage) on chest radiograph from day 1 (randomization) to day 7
* To determine the change on inflammatory markers (WBC/CRP) from day 1 (randomization) to day 7
* To determine the outcome :

  * Length of hospital stay (in days) after randomization for each group
  * The need of surgical intervention in 30 days
  * Adverse effects following t-PA/DNase and pleural irrigation
  * Mortality rate at 30 days

Study Hypothesis

1. Subjects in the IPFT has more volume of pleural fluid drainage compared with pleural irrigation group
2. Subjects in the IPFT has greater reduction of inflammatory parameters compared with pleural irrigation group
3. Subjects in the IPFT has shorter length of hospital stay compared with pleural irrigation group
4. Subjects in the IPFT has less surgical referral rate compared pleural irrigation group
5. There is no difference of mortality rate between both groups

Subjects with pleural infection (complex parapneumonic effusion or empyema) with poor outflow ≤150cc pleural fluid from chest drain over 24 hours of insertion with standard medical therapy who are eligible for this study will be offered to participate into this study. Patient will be informed that this is an 'off label' drugs and a written informed consent will be obtained.

All patients will undergo chest tube/drain insertion. The decision to insert chest drain, the size of chest drain and when to initiate intrapleural t-PA/DNase is determined by the chest physician.

Ultrasound of thorax and chest radiograph will be performed within 24hours before randomization. Ultrasound of thorax is performed by chest physician with curve probe (ultrasound Mindray, model Z5) for confirmation of complex pleural effusions and chest tube's position. Complex pleural effusion on ultrasound is defined as fibrin strands or septa within the pleural effusion along with presence of loculations in pleural cavity. A baseline chest radiograph will be performed within 24 hours prior to intrapleural fibrinolysis or pleural irrigation to ensure the chest tube position.

Demographic data was collected prior to randomization, which consist of age,gender,ethnicity,BMI,comorbidities. Subjects will be randomized with a block of 4 (using sealed envelope) with random permutations of 2 groups : pleural irrigation group and intrapleural t-PA and DNase.

All patients that prescribed intrapleural t-PA/DNase during the study period will receive a standard dose of medications as below (Appendix 1).

Medication Regimen :

t-PA (Alteplase) 5mg and DNase (Pulmozyme)5mg t-PA (Alteplase) that is available in our pharmacy is 50mg ampoule and DNase (Pulmozyme) is 2.5mg per ampoule The number of installation of intrapleural t-PA/DNase depends on the discretion of the treating physician (at least 6 hours apart between each dose). 5mg of Alteplase (t-PA) and 5mg DNase are diluted in each 50ml of 0.9% sodium chloride solution. t-PA and DNase are not mixed together in one syringe. The detailed method of t-PA/DNase therapy administration is described in Appendix 1. In brief , both medication are administered sequentially which t-PA is first instilled intrapleurally and the chest tube is then clamped for 45 minutes, then unclamped to allow free drainage for 45 minutes. The same procedure is then repeated for DNase. Selection of the timing of treatment and removal of chest tube are depending on the chest physician's judgement.

However, as for patients who were randomized into pleural irrigation group, subjects were administered 250 ml of 0.9% sodium chloride via chest tube a three way tap from a drip stand which were allowed drainage freely over 1 hour. Pleural irrigation will be performed minimum of 3 installations and maximum of 9 installation (3 times per day).

Both groups received standard care of treatment : which includes regular flushing of chest drain to maintain patency using 20mls of normal saline.

The primary outcome was to evaluate the volume of pleural effusion drainage (in mls) 72 hours following randomization. The volume drained measured after subtracting the amount of volume administered as per protocol.

The secondary outcome are measured by the change in the area of pleural opacity in chest x-ray (day 7 post t-PA/DNase compared to baseline), measured as the percentage of the ipsilateral hemithorax occupied by effusion. The area of pleural opacity and the area of the ipsilateral hemithorax will be measured digitally by two radiologists using Horos Project Software, v3.2.1 as described previously in Multicentre Intrapleural Sepsis Trial 2 (MIST-2)

Other outcomes that will be monitored include :

1. Inflammatory markers including serum C-reactive protein (CRP) & white blood count
2. Length of hospital stay in days
3. The need of surgical intervention within 30 days
4. Adverse effects :

   1. Chest pain required escalation of analgesics
   2. Systemic bleeding
   3. Pleural bleeding

During any point of treatment subjects will be allowed to cross-over and analysis will be done as per intention to treat. Subjects in the pleural irrigation group may be switched to IPFT group if there is poor response to treatment (poor drainage of effusion), or adverse effects of irrigation as per clinician's judgement. On the contrary, subjects in the IPFT group may be switched to pleural irrigation group if patient developed any adverse effects of IPFT (e.g hemothorax,haemoptysis). Those who failed both treatment will be referred for surgical intervention

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with aged ≥ 18 years old 2. Patients with pleural infection (complex parapneumonic effusion or empyema) with poor pleural fluid drainage of ≤ 150 ml after 24H of insertion of chest drain 3. Clinical features consistent with pleural infection ; fulfilling ≥ 2 of the following characteristics : i) Clinical evidence of infection such as fever and or elevated C-reactive protein (CRP) or total white blood count (TWBC) ii) Complex pleural effusion proven by thoracic ultrasound is defined as presence of fibrin strands or septations within pleural cavity iii) Pleural fluid that fulfil at least one of the characteristic :

* frank pus,
* exudative type of pleural effusion (according to light's criteria)
* gram stain or culture positive
* lactate dehydrogenase (LDH) > 900U/L
* Acidic with ph < 7.2
* glucose level < 3.3 mmol/L

Exclusion Criteria:

1. Refusal to participate
2. Known allergy to t-PA or DNase
3. Acute stroke
4. Significant bleeding diathesis/ active gastrointestinal bleed
5. Major surgery in the previous 5 days
6. Previous pneumonectomy on the infected side
7. Bronchopleural fistula
8. Pregnancy
9. Coagulapathy (INR > 2, APTT > 100)
10. Platelet count < 50000 cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
to evaluate the volume of pleural effusion drainage (in mls) 72 hours following randomization. | 72 hours
  The net volume of pleural effusion drained measured after subtracting the amount of volume administered as per protocol.

SECONDARY OUTCOMES:
To measure the change in the area of pleural opacity in chest x-ray compared to baseline | Day 7
  measured as the percentage of the ipsilateral hemithorax occupied by effusion. The area of pleural opacity and the area of the ipsilateral hemithorax will be measured digitally by two radiologists using Horos Project Software, v3.2.1 as described previously in Multicentre Intrapleural Sepsis Trial 2 (MIST-2)
Changes in Inflammatory markers including serum C-reactive protein (CRP) & white blood count | Day 7
  reduction of inflammatory markers trend
Length of hospitalization | through admission (up to 30 days)
  measured in days
adverse events post therapy | Day 7
  pain, bleeding events, hemodynamically stability
the need for surgical referral | throughout admission up to 30 days
  If failed intrapleural fibrinolytic or pleural irrigation (Discretion of treating physician)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS (IIUM), Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT05903417/Prot_SAP_ICF_000.pdf